CLINICAL TRIAL: NCT02760186
Title: Effect of High Altitude Exposure, Acclimatization and Re-exposure on Lung Water Content by Ultrasound
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: REB15-2709_V5
Record Dates: First submitted 2016-04-12; First posted 2016-05-03 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Effect of High Altitude

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Altitude Exposure (Experimental): Acute high altitude exposure followed by 7 day acclimatization and reexposure after 7 days at low altitude
  Interventions: Procedure: Altitude Exposure

INTERVENTIONS:
Procedure: Altitude Exposure — Altitude Exposure

SUMMARY:
Prospective interventional trial in lowlanders evaluating effect of acute exposure, acclimatization and re-exposure to high altitude.

DETAILED DESCRIPTION:
Low altitude baseline measurements will be performed in Santiago de Chile, 520 m, over the course of 3 days. Participants will then travel by commercial airline (5 h flight) and by bus (3 h ride) to the Atacama large Millimeter Array (ALMA) base camp located at 2900 m near San Pedro de Atacama, northern Chile. Participants will stay there for the next 7 nights and they will be spend the days (6-8 h daily) at the telescope station at 5050 m while undergoing physiological testing. Daily transports from 2900 to 5050 m will be by car (1 h ride, one way). After the first 7 day altitude sojourn participants will return to the Santiago area (520 m) for a 7 day recovery period.

A second altitude sojourn cycle with an identical schedule as the one described above and a final low altitude stay of 3 days will follow.

Measurements on study subjects will be performed at baseline (lowland, Santiago de Chile), then at 2nd day of altitude exposure and 7th day at altitude before returning to lowland; those are repeated in the second altitude sojourn cycle. Measurements will be conducted by qualified specialists using a portable ultrasound device.

ELIGIBILITY:
Inclusion Criteria:

* Born, raised and currently living <800m
* No overnight stay at altitudes > 1500m 4 weeks before the study

Exclusion Criteria:

* Previous altitude intolerance to altitude <3000m
* Pregnancy
* Health impairment, which requires regular treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-03; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
ultrasound lung comets | change from lowland baseline at 520m, day 2 and first sojourn at 5050 m, day 2

SECONDARY OUTCOMES:
ultrasound lung comets | first sojourn at 5050 m, 7; second sojourn at 5050m, day 2, 7

CONTACTS AND LOCATIONS:
Overall Officials: Konrad E Bloch, MD, Study Chair — University of Zurich
Locations (1):
- Switzerland, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided